CLINICAL TRIAL: NCT04745052
Title: Establishment and Validation of a Predictive Model for Hemorrhage After Intravenous Thrombolysis in Acute Ischemic Stroke
Brief Title: Establishment and Validation of a Predictive Model for Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20203357004
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
Keywords: Hemorrhagic transformation; Thrombolysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke: The first is to verify the application effect of intravenous thrombolytic hemorrhage prediction models (HAT, SIT-sICH, THRIVE) in the population of acute ischemic stroke in Guangdong Province, and verify the clinical application effects of existing prediction models. Secondly, analyze the predictive value of clinical indicators, optimize HAT, SIT-sICH, and THRIVE scores, construct an improved HT prediction model, and optimize and improve the existing prediction model. The third is to apply the improved HT prediction model to the clinic, collect clinical data prospectively, evaluate the prediction effect of the model, and evaluate the clinical application effect of the improved prediction model.
  Interventions: Other: Clinical observation index

INTERVENTIONS:
Other: Clinical observation index — The first is to verify the application effect of intravenous thrombolytic hemorrhage prediction models (HAT, SIT-sICH, THRIVE) in the population of acute ischemic stroke in Guangdong Province, and verify the clinical application effects of existing prediction models. Secondly, analyze the predictive value of clinical indicators, optimize HAT, SIT-sICH, and THRIVE scores, construct an improved HT prediction model, and optimize and improve the existing prediction model. The third is to apply the improved HT prediction model to the clinic, collect clinical data prospectively, evaluate the prediction effect of the model, and evaluate the clinical application effect of the improved prediction model.

SUMMARY:
Background: Patients with acute ischemic stroke (AIS) are at risk of hemorrhagic transformation (HT) after intravenous thrombolysis. Although there is a risk assessment model for hemorrhagic transformation after thrombolysis, there is no evidence of clinical application in the population of Guangdong Province. .

Purpose: To verify the clinical application effect of the existing risk assessment model for hemorrhage transformation after thrombolysis in the local population; to improve the existing prediction model and verify the predictive value of HT after intravenous thrombolysis.

Methods: (1) Continuously collect AIS patients who received intravenous thrombolysis in our hospital from January 2014 to December 2020 to verify the clinical application effects of three existing models (HAT, SIT-sICH, THRIVE) on bleeding transformation. Collect baseline and bleeding transformation information within 7 days after thrombolysis, and use ROC curve, calibration curve, sensitivity and specificity to evaluate the prediction effect. A logistic regression model was used to construct an improved HT prediction model based on the AIC principle; (2) Continuous collection of AIS patients who received intravenous thrombolysis in two local hospitals from January 2021 to December 2022 for internal and external verification.

Expected results: (1) Evaluate the clinical application value of the existing prediction model in local AIS patients with intravenous thrombolysis; (2) Develop a modified risk assessment model suitable for hemorrhage transformation after intravenous thrombolysis in AIS patients in Guangdong area, and evaluate the risk early Provide guarantee for clinical diagnosis and treatment.

DETAILED DESCRIPTION:
This study has two main parts. The first part is to verify and optimize the clinical application effect of the existing prediction model. The clinical data of the acute ischemic stroke intravenous thrombolytic population is collected retrospectively, mainly including baseline indicators and 7 days after thrombolysis Internal bleeding, based on the existing prediction models (HAT, SIT-sICH, THRIVE), calculate the prediction probability, and compare it with the actual bleeding situation, evaluate the clinical application effect of the prediction model, use ROC curve, calibration curve, sensitivity and Evaluation of indicators such as specificity. Using retrospective data, using multivariate logistic regression to analyze the predictive value of baseline clinical indicators, screening risk factors, and optimizing the HAT, SIT-sICH, and THRIVE prediction models. The logistic regression model is used to construct an improved HT prediction model based on the AIC principle; the method of model comparison is used to combine the clinical significance of the indicators to complete the construction of the prediction model. The second part is to evaluate the clinical application effect of the improved prediction model, and prospectively collect clinical data of AIS patients undergoing intravenous thrombolysis in Shenzhen Second People's Hospital, Shenzhen Longhua District People's Hospital, including general demographic data and laboratory tests Baseline indicators such as imaging examinations, bleeding within 7 days after thrombolysis, etc., were used to verify the improved HT prediction model using ROC curve, calibration curve, sensitivity and specificity, and external verification was performed to evaluate the prediction effect of the model.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Onset time <4.5 hours;
3. Meet the diagnostic criteria of the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018, and have been examined by plain CT/MRI of the head, and hemorrhagic stroke is excluded by head CT;
4. AIS patients receiving intravenous thrombolysis.

Exclusion Criteria:

1. The main clinical data is incomplete;
2. Patients treated by intraarterial thrombolysis or interventional thrombectomy;
3. Patients with transient ischemic attack;
4. Those who refuse to participate in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke in Shenzhen Second People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Build HT prediction model | March 1, 2021 to March 1, 2022
  Collect baseline and bleeding transformation information within 7 days after thrombolysis, and use ROC curve, calibration curve, sensitivity and specificity to evaluate the prediction effect. Use logistic regression model to build an improved HT prediction model based on AIC principles

CONTACTS AND LOCATIONS:
Overall Officials: Xie Xiaohua, master, Principal Investigator — Director of Nursing
Locations (2):
- China (2):
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - China, Guandong, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided